CLINICAL TRIAL: NCT02333734
Title: Investigation of the Effect of 8-week Controlled High Intense Interval Training in Type 2 Diabetic Patients
Acronym: DIATRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Per Bendix Jeppesen, Research Associate Prof. PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: T2D-training; Aarhus University (Other: Aarhus University)
Record Dates: First submitted 2014-07-08; First posted 2015-01-07 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Interval training; Insulin resistance; fat metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Type 2 diabetic subjects (Experimental): Type 2 diabetic subjects physical training (interval training 3 times at week) in a period of 8 weeks.
  Interventions: Other: Physical training
- Healthy subjects (Experimental): Healthy subjects physical training (interval training 3 times at week) in a period of 8 weeks.
  Interventions: Other: Physical training

INTERVENTIONS:
Other: Physical training — Performed supervised high intensity interval training 3 times a week over 8 weeks on a bicycle ergometer (with watt meter). During the training period, the trainee individually established program, each time with 10 × 60 sec. workout (interspersed with 60 sec. break) corresponding to a force which during the test cycle induces ~ 90% of the maximum heart rate. The time spent per session is expected to last ~ 25 minutes.

SUMMARY:
The overall objective of this study is to examine the blood flow in the thigh muscles and sugar metabolism before and after 8 weeks of high intensity interval training (HIIT) on a bicycle ergometer in patients with type 2 diabetes (T2D) and matched controls. The following parameters are included in the assessment:

* Sugar Metabolism
* Muscle and fat mass
* The blood flow at rest around the thigh muscles
* Oxygen uptake test on a bicycle ergometer and 5 km time trial

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) can be defined as a bihormonal metabolic disorder characterised by insufficient insulin secretion and abnormal glucagon secretion. It is however well established that physical activity per se improves glucose and may postpone or even slow down in the diabetic population. Glycaemic control may be improved more by high intensity interval training than by intensities from existing recommended guidelines. Additionally, there seems to be accumulating evidence that high intensity interval training induces increased overall fat and abdominal fat mass loss as opposed to traditional continuous endurance training Therefore we hypothesise that 3 weekly sessions of high intensity interval training (10×60 sec. at an intensity inducing 90% of maximal heart frequency with a recovery of 60 sec. between each bout) over 8 weeks improves overall glycaemic control (glucose, insulin and glucagon), inflammatory status (interleukins, cytokines, chemokines and cell adhesion molecules) and blood flow (NO and PGI2 vasodilatory capabilities).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes or matched healthy controls. T2D subject only : HbA1c > 7,3. All subjects have an age between 40-65 years and a body mass index between 25-40 kg/m2. Both genders is allowed

Exclusion Criteria:

* Severe diseases /immobility

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Oral Glucose tolerance test (OGTT) | baseline and 8 weeks
  Change from baseline and 8 weeks in glucose/insulin response from a 2.5 hours oral glucose tolerance test (iAUC) after 8 weeks training

SECONDARY OUTCOMES:
Physical fitness | baseline and 8 weeks
  Change from baseline and after 8 weeks in physical fitness level (mL/min x kg) measured with submaximal test using a bicycle ergometer after 8 weeks interval training .

OTHER OUTCOMES:
Muscle and fat mass | baseline and 8 weeks
  Change from baseline and 8 weeks in Muscle and fat mass (DEXA Scan)
blood flow | baseline and 8 weeks
  Change from baseline and 8 weeks in blood flow at rest around the thigh muscles (Ultra Sound technic)

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus Universityhospital, Aarhus University, Aarhus C, Denmark

REFERENCES:
- [Derived] Madsen SM, Thorup AC, Overgaard K, Jeppesen PB. High Intensity Interval Training Improves Glycaemic Control and Pancreatic beta Cell Function of Type 2 Diabetes Patients. PLoS One. 2015 Aug 10;10(8):e0133286. doi: 10.1371/journal.pone.0133286. eCollection 2015. PMID 26258597